CLINICAL TRIAL: NCT05956314
Title: Phase 1b, Open Label Study to Evaluate the Safety, Tolerability, and Efficacy of a 1% Topical Formulation of KM-001 for the Treatment of Type I Punctate Palmoplantar Keratoderma or Pachyonychia Congenita
Brief Title: Assessment of KM-001 - Safety, Tolerability, and Efficacy in Patients With PPPK1 or PC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kamari Pharma Ltd (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KM001-B1B
Record Dates: First submitted 2023-06-14; First posted 2023-07-21 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-04

CONDITIONS: Punctate Palmoplantar Keratoderma Type 1; Pachyonychia Congenita
MeSH Terms: conditions — Keratosis palmoplantaris papulosa; Pachyonychia Congenita | interventions — Therapeutics; Physical Examination; Vital Signs; Hematologic Tests; Urinalysis; Pain Measurement

STUDY DESIGN:
Intervention Model Description: In this phase 1b, open label trial, 2 arms will be treated twice daily with 1% topical KM-001 (2 feet):
  1. Arm 1: up to 11 eligible patients.
  2. Arm 2: up to 7 eligible patients. During active treatment, safety, tolerability, efficacy, and PK assessments will be performed. Four (4) weeks after the end of active treatment, patients will return to the clinic for additional safety, efficacy, and PK assessments.
  Safety, tolerability, and efficacy parameters will be assessed during in-clinic visits as follow:
  For both cohorts: Screening, Enrolment, Days 7, 28, 42, 63.
  Additionally:
  For arm 1: Day 84 [end of treatment], 112 [End of Study] For arm 2: day 84, 112 [EoT] and 140 EoS] post first investigational medicinal product (IMP) administration.
  Safety and treatment compliance assessment will be done by phone calls on - Cohort 1: Days 14, 49, 70, and 98 (follow-up); Cohort 2: Days 14, 49, 70, 98, and 126 (follow-up).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KM-001 cream 1% 12 weeks treatment. (Experimental): KM-001 1% cream will be applied to the affected area, twice daily for 12 consecutive weeks.
  KM-001 will be supplied in glass jars (30 g) and will be provided to patients with spatulas and polyethylene gloves.
  Interventions: Drug: KM-001 cream 1% 12 weeks treatment.; Diagnostic Test: Physical Examination; Diagnostic Test: Vital Signs; Diagnostic Test: Serum chemistry; Diagnostic Test: Hematology; Diagnostic Test: Serology; Diagnostic Test: Urinalysis; Diagnostic Test: ECG test; Diagnostic Test: Pharmacokinetics Assessments; Diagnostic Test: Clinical global impression of severity (CGI-S); Diagnostic Test: Visual Analogue Scale (VAS) pain scale; Diagnostic Test: Peak pruritus-numerical rating scale (PP-NRS); Diagnostic Test: Patient global impression of change (PGI-C) scoring; Diagnostic Test: Patient global impression of severity (PGI-S) scoring; Diagnostic Test: Lesion photography
- KM-001 cream 1% 16 weeks treatment. (Experimental): KM-001 1% cream will be applied to the affected area, twice daily for 16 consecutive weeks.
  KM-001 will be supplied in glass jars (30 g) and will be provided to patients with spatulas and polyethylene gloves.
  Interventions: Diagnostic Test: Physical Examination; Diagnostic Test: Vital Signs; Diagnostic Test: Serum chemistry; Diagnostic Test: Hematology; Diagnostic Test: Serology; Diagnostic Test: Urinalysis; Diagnostic Test: ECG test; Diagnostic Test: Pharmacokinetics Assessments; Diagnostic Test: Clinical global impression of severity (CGI-S); Diagnostic Test: Visual Analogue Scale (VAS) pain scale; Diagnostic Test: Peak pruritus-numerical rating scale (PP-NRS); Diagnostic Test: Patient global impression of change (PGI-C) scoring; Diagnostic Test: Patient global impression of severity (PGI-S) scoring; Diagnostic Test: Lesion photography; Drug: KM-001 cream 1% 16 weeks treatment.

INTERVENTIONS:
Drug: KM-001 cream 1% 12 weeks treatment. — KM-001 1% will be supplied in glass jars (30 ml) and will be provided to patients with spatulas and polyethylene gloves on all the clinical visits. The patient will use IMP twice a day for 84 days. IMP will be applied on the plantar surfaces.
  Other Names: Experimental drug administration-cohort 1
  Arms: KM-001 cream 1% 12 weeks treatment.
Diagnostic Test: Physical Examination — A complete physical examination will be performed as follows at screening and baseline, abbreviated after that (i.e., on Days 7, 28, 42, 63, 84, 112, 140, and at ET visit - where applicable, per cohort):
  * The complete physical examination will cover a careful assessment of all body systems, including the head, eyes, ears, nose, and throat and the respiratory, cardiovascular, gastrointestinal (GI), musculoskeletal, neurological, dermatological, hematologic/lymphatic, and endocrine systems. Particular attention will be placed on the areas affected by the disease.
  * Symptom-directed physical examinations will be performed at all other trial visits.
  * Height and weight measurement will be performed at screening only. An abbreviated examination including a comprehensive skin examination.
Diagnostic Test: Vital Signs — Vital sign measurements (oral body temperature, pulse, and resting systolic and diastolic blood pressure) will be measured at screening, on Days 1, 7, 28, 42, 63, 84, 112, 140, and at ET visit - where applicable, per cohort. Vital signs will be measured in supine position after at least 5 minutes of rest.
Diagnostic Test: Serum chemistry — Approx. 5 mL whole blood will be collected after an ≥8 h fast for serum biochemistry assessments during screening, and on Days 1 (baseline), 7, 84 112, 140 or at an ET visit - where applicable, per cohort. Serum chemistry will include assessments of total and direct bilirubin, ALT, AST, gamma-glutamyl transferase (GGT), alkaline phosphatase, glucose (fasting), sodium, potassium, blood urea nitrogen (BUN/Urea), creatinine, chloride, calcium, uric acid, albumin, and total protein.
Diagnostic Test: Hematology — Approx. 5 mL whole blood will be collected for complete blood count (CBC) during screening, and on Days 1 (baseline), 7, 84, 112, 140 or at an ET visit - where applicable, per cohort. The CBC assessments will include red blood cells (RBC), haemoglobin, haematocrit, reticulocyte count, platelet count, mean corpuscular haemoglobin (MCH), mean platelet volume (MCV), white blood cells (WBC), neutrophils (absolute [abs.]), lymphocytes (abs.), monocytes (abs.), eosinophils (abs.), and basophils (abs.).
Diagnostic Test: Serology — Approx. 5 mL whole blood will be collected for serology assessments during screening. Serology will include HbsAg, HbcAb, hepatitis C antibody, and HIV antibody.
Diagnostic Test: Urinalysis — General urinalysis will be performed, by dipstick, during screening, and on Days 1 (baseline), 7, and 84, 112, and 140, or at an ET visit - where applicable, per cohort. At least 7 to 10 mL of urine will be collected. Urinalysis will include pH, specific gravity, blood, nitrites, glucose, ketones, protein, bilirubin, urobilinogen, and leukocytes. A microscopic examination of the urine will be performed only if clinically indicated.
Diagnostic Test: ECG test — A 12-lead, resting, ECG will be taken for each patient at screening, on Days 1 (baseline), 84, 112, and at day 140 (for Cohort 2), or at an ET visit - Where applicable. The measurement will be taken after the patient has been supine for at least 5 min. At minimum, the following ECG parameters will be recorded: heart rate (HR), PR, QT, and QTc interval and QRS complex. The report will be printed out and signed by the investigator, who will record in the eCRF whether it is normal, abnormal but not clinically significant, or abnormal AND clinically significant. In the latter case the eligibility of the patients will be reviewed.
Diagnostic Test: Pharmacokinetics Assessments — Blood samples for PK will be collected during screening (Days -14 to 0) at any time during the visit, or on Day 1 (up to 30 minutes prior to the first dose, if not performed during Screening) and on Day 7 and at End of Treatment (EoT, Cohort 1: Day 84; Cohort 2: Day 112) up to 30 minutes pre-dose and at 1 h, 2 h, 3 h, 6 h (+15 min) post-dose, on Days 28, 42, and 84 (for Cohort 2): 1 sample after the first dose, before the second dose, as late as possible in the visit, at End of Study (EoS, Cohort 1: Day 112; Cohort 2: Day 140), or at an ET visit: at any time during the visit.
  * Altogether up to 15 samples, and approx. 30 mL of blood will be drawn for PK at screening or Day 1 and on Days 7, 28, 42, 84, EoT (84/112), and EoS (112/140), or at an ET visit, if applicable.
  * Overall, up to a total of 85 mL of blood will be drawn during the trial for blood and PK assessments per patient in Cohort 1, and 95 mL of blood per patient in Cohort 2.
Diagnostic Test: Clinical global impression of severity (CGI-S) — Lesions severity will be assessed using the CGI-S scale, which is a 5-point scale (from 0= "none" to 4= "very severe") modified from Busner et al. 2007 (30) by the investigator during screening and on Days 1 (baseline, prior to first dosing), 7, 28, 42, 63, 84, 112, 140, and at ET visit - where applicable, per cohort).
  The clinician scoring takes into account all available information, including a knowledge of the patient's history, psychosocial circumstances, symptoms (pain), behaviour, and the impact of the symptoms on the patient's ability to function (ability to walk). investigators will complete the CGI-S at various timepoints based on the question. "Please choose the response that best describes your assessment of the disease severity, based upon the totality of information available to you"
Diagnostic Test: Visual Analogue Scale (VAS) pain scale — The patient will enter the PPPK- or PC-related pain score (not any pain) using a VAS pain scale in the patient-reported diary, on a weekly basis starting on Day 1 through ET visit, prior to the second administration of the IMP (evening dose) at the same time every time (±1 hour) except for Day 1 (Visit 2, in-clinic visit), where the assessment will be performed pre-dose during the visit.
  The score will be collected on every in-clinic visit during the treatment and follow up periods (Days 1, 7, 28, 42, 63, 84, 112, 140, and at an ET visit - where applicable, per cohort).
  The following parameter will be evaluated on a VAS from 0 (no pain) to 100 (severe intolerable pain) based on the question:
  "How was your worst pain intensity in the past 24 hours?"
Diagnostic Test: Peak pruritus-numerical rating scale (PP-NRS) — The peak pruritus severity will be assessed using the PP-NRS, an 11-point scale from 0 (no itch) to 10 (worst imaginable itch). The PP-NRS will be entered by the patients on a weekly basis starting on Day 1 through ET visit, preferably after the evening dose, at the same time every time (±1 hour) except for Day 1 (Visit 2, in-clinic visit), where the assessment will be performed pre-dose during the visit.
  The scores will be collected on every in-clinic visit during the treatment and follow up periods (Days 1, 7, 28, 42, 63, 84, 112, and 140, or at an ET visit - where applicable, per cohort).
  The PP-NRS was designed to measure peak pruritus, or "worst" itch, over the previous 24 hours based on the following question: "On scale from 0 (no itch) to 10 (worst imaginable itch) how was your worst itch in the past 24 hours?"
Diagnostic Test: Patient global impression of change (PGI-C) scoring — The PGI will be evaluated on Days 1, 7, 28, 42, 63, 84, 112, and 140, or at an ET visit - where applicable, per cohort.
  The PGI-C will be evaluated using a 7-point scale from 1 (very much improved) to 7 (very much worse) as follows:
  Since the start of the trial, my overall status has:
  from, 1= "very much improved" to 7= "very much worse"
Diagnostic Test: Patient global impression of severity (PGI-S) scoring — The PGI will be evaluated on Days 1, 7, 28, 42, 63, 84, 112, and 140, or at an ET visit - where applicable, per cohort.
  The PGI-S will be evaluated using a 5-point scale from 1 (none) to 5 (very severe) as follows:
  Please rate the severity of your disease right now, from 1= "none" to 5= "very severe"
Diagnostic Test: Lesion photography — High quality photographic documentation of the treated lesions will be performed during Screening and on Days 1, 7, 42, 63, 84, 112, and 140, or at an ET visit before treatment - where applicable, per cohort.
  The photographs will be taken under standardised conditions, using imitoMeasure (Ⓒ imito AG 2016-2022).
Drug: KM-001 cream 1% 16 weeks treatment. — KM-001 1% will be supplied in glass jars (30 ml) and will be provided to patients with spatulas and polyethylene gloves on all the clinical visits. The patient will use IMP twice a day for 112 days. IMP will be applied on the plantar surfaces.
  Other Names: Experimental drug administration-cohort 2
  Arms: KM-001 cream 1% 16 weeks treatment.

SUMMARY:
This Phase 1b, open-label, single-center, prospective trial will be assessing the safety, tolerability, and efficacy of topical KM-001 1% in patients with PPPK1 or PC diseases. In this study 2 cohorts will be recruited:

1. Cohort 1: up to 11 eligible patients, will be enrolled to be treated twice daily, for 12 weeks, with 1% topical KM-001, on the plantar surfaces (2 feet).
2. Cohort 2: up to 8 eligible patients, will be enrolled to be treated twice daily, for 16 weeks, with 1% topical KM-001, on the plantar surfaces (2 feet).

Safety (AEs, blood work [at specific visits], vital signs), tolerability, and efficacy parameters (overall lesion improvement) will be assessed during in-clinic visits (Cohort 1: during Screening, Enrolment, and on Days 7, 28, 42, 63, 84 [end of treatment, EoT], 112 [End of Study, EoS] post first investigational medicinal product (IMP) administration; Cohort 2: during Screening, Enrolment, and on Days 7, 28, 42, 63, 84, 112 [EoT], 140 [EoS] post first investigational medicinal product (IMP) administration).

PK samples will be collected to assess plasma levels of KM-001 on

* Screening (Day -14 to -0): any time during the visit. (or on Day 1 up to 30 minutes pre-dose if missed during Screening)
* Day 7 and at EoT (Cohort 1: Day 84; Cohort 2: Day 112) up to 30 minutes pre-dose, and at 1 h, 2 h, 3 h, 6 h (+15 min) post-dose
* Days 28, 42 for both Cohorts, and Day 84 for Cohort 2: 1 sample after the first dose, before the second dose, as late as possible in the visit.
* End of Study (EoS, Day 112 (Cohort 1) or Day 140 (cohort 2)), or at Early Termination (ET): at any time during the visit.

The patient will complete a patient-reported diary, consisting of treatment compliance and self-assessments for efficacy.

Follow up- 2 weeks after EoT by phone call, and 4 weeks after EoT in clinic visit.

DETAILED DESCRIPTION:
The palmoplantar keratoderma (PPK) group of skin disorders results from various mutations in several epidermal genes and is characterized by thickening of the skin on the palms and soles.

Punctate palmoplantar keratoderma (PPKP1) is a rare autosomal, dominant, inherited skin disease characterized by bilateral asymptomatic, tiny, hyperkeratotic punctate papules and plaques on the palmoplantar surface.

Pachyonychia congenita (PC) is a rare group of autosomal dominant skin disorders that are caused by a mutation in one of five different keratin genes. PC is often associated with thickened toenails, plantar keratoderma, and plantar pain. Its manifestations include bilateral PPK on palms and soles pattern with sharp margins and a yellow tone.

A common characteristic of these skin diseases is the impaired differentiation of keratinocytes, often caused by defective calcium homeostasis. Normal calcium homeostasis is regulated by calcium ion channels, including the transient receptor potential cation channel subfamily V, member 3 (TRPV3), which has been implicated in regulation of keratinocyte proliferation, differentiation, and apoptosis. As a result, it has been suggested as a drug target for a variety of dermatological conditions and itch. It has therefore been suggested that inhibition of TRPV3 by specific antagonists can address the above-mentioned conditions.KM-001, developed by Kamari Pharma, is a potent and selective TRPV3 antagonist. Kamari has demonstrated that KM-001 reduces Ca+2flux in keratinocytes and decreases cell proliferation accompanied by normalization of keratinocyte differentiation markers. Efficacy was demonstrated in in vivo studies, using the DS-Nh mice model, where it was able to normalize epidermal hyperkeratosis. In addition, the compound significantly reduced pruritus which is characteristic of this model and of many types of PPK.

KM-001 topical formulation demonstrates favorable safety profile in rodents and minipigs and significant efficacy in animal models.

ELIGIBILITY:
Inclusion Criteria:

1. Read, understood, and signed an informed consent form (ICF) before any investigational procedure(s) are performed.
2. Male and female and aged 18 - 75 years (inclusive) at the time of screening.
3. Clinical diagnosis of:

   • Punctate palmoplantar keratoderma type I disease with confirmed heterozygous mutation in AAGAB gene.

   OR

   • PC with confirmed heterozygous mutation in either KRT16, KRT17, KRT6A, KRT6B or KRT6C mutations.
4. The target treatment region is 0.5% to 4% BSA including target lesion.
5. CGI-S score (as assessed by the CI at the screening visit) of ≥2.
6. Female patients of childbearing potential1 must use a highly effective birth control method2 (failure rate ˂1% per year when used consistently and correctly) (28) throughout the trial and for at least 4 weeks after last application of IMP.

In addition to the hormonal contraception, female patients must agree to use a supplemental barrier method during intercourse with a male partner (i.e., male condom) throughout the trial and for at least 4 weeks after last application of IMP.

Female patients must be having regular menstrual periods (interval of 21 to 35 days, duration of 2 to 7 days for several months) at the baseline visit (as reported by the patient); exception: patients using hormonal contraceptives that preclude regular menstrual periods, menopausal or hysterectomised patients.

A male patient with a pregnant or non-pregnant female partner of childbearing potential1 must use adequate contraceptive methods (adequate contraceptive measures as required by local regulation or practice; as a minimum, the male patient must agree to use condom during treatment and until the end of relevant systemic exposure in the male patient (7 days post-treatment).

1. A female patient is considered of childbearing potential, i.e., fertile, following menarche and until becoming postmenopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy. A postmenopausal state is defined as no menses for at least 12 months without an alternative medical cause prior to screening (28).
2. Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal) or progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable) 28 days prior to screening, bilateral tubal occlusion, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), vasectomised/permanently sterile by bilateral orchidectomy partner (given that the partner is the sole sexual partner and has received medical assessment of the surgical success), or sexual abstinence (refraining from heterosexual intercourse during the entire trial/treatment period of risk associated with the IMPs) (28). This period of contraception should be extended for at least 4 weeks after last application of IMP.

7. Female patients must refrain from donating eggs throughout the trial and for 4 weeks after the last IMP administration.

Male patients must refrain from sperm donation throughout the trial and for 7 days after the last IMP administration.

8. Female patients of non-childbearing potential must meet 1 of the following criteria:

1. Absence of menstrual bleeding for 1 year prior to screening without any other medical reason.
2. Documented hysterectomy or bilateral oophorectomy at least 3 months before the trial.

   9. Patient is willing and able to comply with all the time commitments and procedural requirements of the protocol.

   Exclusion Criteria:
   1. History of drug or alcohol abuse in the past 2 years.
   2. Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine).
   3. Positive hepatitis B surface antigen [HbsAg], hepatitis B core antibody [HbcAb], hepatitis C antibody, or human immunodeficiency virus (HIV) antibody serology results at the screening visit.
   4. Known hypersensitivity or any suspected cross-allergy to the API and/or excipients.
   5. Any medical or active psychological condition or any clinically relevant laboratory abnormalities, such as, but not limited, to elevated alanine aminotransferase (ALT) or aspartate aminotransferase (AST) (>3 × upper limit of normal [ULN]) in combination with elevated bilirubin (>2 × ULN), at the screening/baseline visit.
   6. Planned or expected major surgical procedure during the clinical trial.
   7. Patient is unwilling to refrain from using prohibited medications during the clinical trial.
   8. Currently participating or participated in any other clinical trial of an IMP or device, within the past 4 months before the screening visit.
   9. Cutaneous infection or another underlying condition of the skin which may impact the assessments or trial participation.
   10. Cutaneous infection of the area to be treated with IMP within 2 weeks before the screening visit or any infection of treatment area requiring treatment with oral, parenteral antibiotics, antivirals, antiparasitics or antifungals or any topical within 2 weeks before the screening visit.
   11. Pregnant or breastfeeding patient.
   12. Failure to satisfy the investigator of fitness to participate for any other reason.
   13. Having received any of the prohibited treatments in Table 5 within the specified timeframe before the baseline visit.

       -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-11-07 (Actual)

PRIMARY OUTCOMES:
Safety endpoint will be assessed through collection and analysis of adverse events. | Up to 112 days
  Incidence rate of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) grouped by body system up to the patient´s end of trial (Day 112 [Visit 12]) or early termination [ET] visit]).
Safety endpoint-will be assessed by the % of change from normal range in the collection of Hematology- laboratory blood test profile. | Up to 112 days
  Safety will be assessed by the % of change from normal range in clinical Hematology blood test profile from baseline (Day 1) up to day 112.
  Data management team will assess and review the laboratory blood test results (Hematology). Exceptional values above the norm or below the norm indicate an aggravation of the participant's condition.
  The following values will be assessed: WBC (K/µl) and platelet count (K/µl), neutrophils (absolute [abs.])(K/µl), lymphocytes (abs.)(K/µl), monocytes (abs.) (K/µl), eosinophiles (abs.)(K/µl) and basophiles (abs.) (K/µl) and reticulocyte count (K/µl).
Safety endpoint-will be assessed by the % of change from normal range in the collection of MCH result in laboratory blood test. | Up to 112 days
  Safety will be assessed by the % of change from normal range in MCH (pg) blood test result, from baseline (Day 1) up to day 112.
  Data management team will assess and review the MCH lab test results. Exceptional values above the norm or below the norm indicate an aggravation of the participant's condition.
Safety endpoint-will be assessed by the % of change from normal range in the collection of MCV result in laboratory blood test. | Up to 112 days
  Safety will be assessed by the % of change from normal range in MCV(fl) laboratory blood test result, from baseline (Day 1) up to day 112.
  Data management team will assess and review the MCV lab test results. Exceptional values above the norm or below the norm indicate an aggravation of the participant's condition.
Safety endpoint-will be assessed by the % of change from normal range in the collection of haematocrit result in laboratory blood test. | Up to 112 days
  Safety will be assessed by the % of change from normal range in haematocrit (%) laboratory blood test result, from baseline (Day 1) up to day 112.
  Data management team will assess and review the haematocrit lab test results. Exceptional values above the norm or below the norm indicate an aggravation of the participant's condition.
Safety endpoint-will be assessed by the % of change from normal range in the collection of hemoglobin result in laboratory blood test. | Up to 112 days
  Safety will be assessed by the % of change from normal range in hemoglobin (g/dL) laboratory blood test result, from baseline (Day 1) up to day 112.
  Data management team will assess and review the hemoglobin lab test results. Exceptional values above the norm or below the norm indicate an aggravation of the participant's condition.
Safety endpoint-will be assessed by the % of change from normal range in the collection of RBC result in laboratory blood test. | Up to 112 days
  Safety will be assessed by the % of change from normal range in RBC (M/µl) laboratory blood test result, from baseline (Day 1) up to day 112.
  Data management team will assess and review the RBC lab test results. Exceptional values above the norm or below the norm indicate an aggravation of the participant's condition.
Safety endpoint-will be assessed by the % of change from normal range in the collection of Sodium, potassium and chloride results in chemistry laboratory blood test. | Up to 112 days
  Safety will be assessed by the % of change from normal range in chemistry laboratory blood test profile, from baseline (Day 1) up to day 112.
  Data management team will assess and review the chemistry lab test results. Exceptional values above the norm or below the norm indicate an aggravation of the participant's condition.
  The following values will be assessed:
  Sodium (mmol/L), potassium (mmol/L) and chloride (mmol/L).
Safety endpoint-will be assessed by the % of change from normal range in the collection of: Glucose fasting , BUN/Ur, creatinine, bilirubin total and direct, calcium, uric acid, and bilirubin result, in chemistry laboratory blood test. | Up to 112 days
  Safety will be assessed by the % of change from normal range in chemistry laboratory blood test profile, from baseline (Day 1) up to day 112.
  Data management team will assess and review the chemistry lab test results. Exceptional values above the norm or below the norm indicate an aggravation of the participant's condition.
  The following values will be assessed:
  Glucose fasting (mg/dL), BUN/Ur (mg/dL), creatinine (mg/dL), bilirubin total (mg/dL) and direct (mg/dL), calcium (mg/dL), uric acid (mg/dL), and bilirubin (mg/dL).
Safety endpoint-will be assessed by the % of change from normal range in the collection of Alkaline phosphatase, AST, ALT and GGT result in chemistry- laboratory blood test. | Up to 112 days
  Safety will be assessed by the % of change from normal range in chemistry laboratory blood test profile, from baseline (Day 1) up to day 112.
  Data management team will assess and review the chemistry lab test results. Exceptional values above the norm or below the norm indicate an aggravation of the participant's condition.
  The following values will be assessed:
  Alkaline phosphatase (U/L), AST (U/L), ALT (U/L) and GGT (U/L).
Safety endpoint-will be assessed by the % of change from normal range in the collection of Albumin and total protein result in chemistry- laboratory blood test. | Up to 112 days
  Safety will be assessed by the % of change from normal range in chemistry blood test profile, from baseline (Day 1) up to day 112.
  Data management team will assess and review the chemistry lab test results. Exceptional values above the norm or below the norm indicate an aggravation of the participant's condition.
  The following values will be assessed:
  Albumin (g/dL) and total protein (g/dL).
Safety endpoint-will be assessed by the % of change from normal range in the collection of Serology -in laboratory blood test profile. | Up to 112 days
  Safety will be assessed by the % of change from normal range in serology clinical blood test profile, from baseline (Day 1) up to Day 112.
  Data management team will assess and review the serology lab test results. Exceptional values above the norm or below the norm indicate an aggravation of the participant's condition.
  The following values will be assessed:
  HBsAg (positive/negative), HBcAb (positive/negative), hepatitis C antibody (positive/negative), or HIV antibody (positive/negative).
Safety endpoint-will be assessed by the % of change from normal range in the collection of urine laboratory profile. | Up to 112 days
  Safety will be assessed by the % of change in clinical urine laboratory profile from baseline (Day 1) up to Day 112.
  Data management team will assess and review the urine lab test results. Exceptional values above the norm or below the norm indicate an aggravation of the participant's condition.
  the following values will be assessed: Glucose (mg/dl), protein (mg/ml),urobilinogen (mg/ml) and ketones (mg/ml).
Safety endpoint-will be assessed by the % of change from normal range in the collection of Specific gravity , pH, blood and nitrites result in urine laboratory profile. | Up to 112 days
  Safety will be assessed by the % of change in clinical urine laboratory profile from baseline (Day 1) up to Day 112.
  Data management team will assess and review the urine lab test results. Exceptional values above the norm or below the norm indicate an aggravation of the participant's condition.
  The following values will be assessed:
  Specific gravity , pH, blood and nitrites.
Safety endpoint-Mean change in body temperature measurement from baseline. | Up to 112 days
  Mean changes in body temperature from baseline (Day 1) up to Day 112.
Safety endpoint-Mean change in pulse measurement from baseline. | Up to 112 days
  Mean changes in pulse (unites: beats per minute) measurements from baseline (Day 1)up to Day 112.
Safety endpoint- Mean change in blood pressure measurement from baseline. | Up to 112 days
  Mean changes in blood pressure (systolic and diastolic blood pressure [unites: mm Hg]) measurements from baseline (Day 1) up to Day 112.
Safety endpoint-ECG | Up to 112 days
  Mean changes in ECG parameters from baseline (Day 1) up to Day 112. the following ECG parameters will be recorded: heart rate (HR), PR, QT, and QTC interval and QRS complex.

SECONDARY OUTCOMES:
Efficacy end point - will be assessed by Clinical global impression of severity (CGI-S) questionaries | Up to 84 days
  Percent responders in CGI-S scale (0= "none" to 4= "very severe") on Day 84 [Visit 10, EoT] compared to baseline (Day 1); a responder is defined to have an improvement of at least 2 points in disease severity on Day 84 [Visit 10, EoT] compared to baseline (Day 1).
Efficacy end point - will be assessed by Patient global impression of change (PGI-S) questionaries | Up to 84 days
  Mean change from baseline (Day 1 [Visit 2] to Day 84 [Visit 10, EoT]) in PGI-S. scale:
  1= "none" 5="very severe"
Efficacy end point - will be assessed by Patient global impression of change (PGI-C) questionaries | Up to 84 days
  Mean change from baseline (Day 1 [Visit 2] to Day 84 [Visit 10, EoT]) in PGI-C. scale:
  1="very much improved" 7="very much worse"

OTHER OUTCOMES:
Exploratory end point- will be assessed by characterize the time to reach Maximum plasma concentration (tmax) of KM-001 | Up to 112 days
  KM-001 plasma levels will be collected at screening (Day -7 to -1, any time during the visit), on Days 7 and 84 (EoT) 1 h, 2 h, 3 h, 6 h (+15 min) post-dose, on Days 28 and 42: 1 sample after the first dose, before the second dose, as late as possible in the visit, on Day 112 and at ET visit: at any time during the visit. The time to reach Maximum plasma concentration (tmax) will be determined.
Exploratory end point- will be assessed by characterize the Area under the plasma concentration versus time curve (AUC) of KM-001 | Up to 112 days
  KM-001 plasma levels will be collected at screening (Day -7 to -1, any time during the visit), on Days 7 and 84 (EoT) 1 h, 2 h, 3 h, 6 h (+15 min) post-dose, on Days 28 and 42: 1 sample after the first dose, before the second dose, as late as possible in the visit, on Day 112 and at ET visit: at any time during the visit. The Area under the plasma concentration versus time curve (AUC) will be determined.
Exploratory end point -will be assess the efficacy of KM-001 1% in pain reduction resulted by Visual analogue scale (VAS) questionnaire. | Up to 84 days
  Mean change from baseline (Day 1 [Visit 2] to Day 84 [Visit 10, EoT]) in pain assessed by VAS score (0= "no pain" to 100= "severe intolerable pain").
Exploratory end point -will be assess the efficacy of KM-001 1% in itch reduction resulted by Peak pruritus-numerical rating scale (PP-NRS) questionnaire. | Up to 84 days
  Itch assessment using the PP-NRS (0= "no itch" to 10= "worst imaginable itch")
Exploratory end point -will be assess the change in the external characteristics of the callus surface using photography and "imitoMeasur" software. | Up to 112 days
  The Changes in the treated callus morphology (Referring to the following parameters: fissuring, neurovascular structures, and erythema around the calluses) will be assessed (decreasing / increasing) using lesions photography. The treated lesions will be photographed using "imitoMeasur" software on Days 1, 7, 28, 42, 63, 84, and 112.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal London Hospital-Clinical Research Facility-11D (11th Floor) Whitechapel, London, E1 1FR,, London, Whitechapel Rd, United Kingdom

IPD SHARING:
Plan to Share IPD: No